CLINICAL TRIAL: NCT05902078
Title: Comparison of the Efficacy and Safety With Eldecalcitol and Calcitriol in Postmenopausal Women With Low Bone Mineral Density or Mild Osteoporosis
Brief Title: Eldecalcitol and Calcitriol in Postmenopausal Women With Low Bone Mineral Density or Mild Osteoporosis
Acronym: EFFECT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Chugai Pharma China Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Zhenlin Zhang, MD, Chief Physician, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023MDEDR0007
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Low Bone Mineral Density; Postmenopausal Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — eldecalcitol; Calcitriol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eldecalcitol (Experimental): Participants receive oral eldecalcitol 0.75μg daily for 12 months
  Interventions: Drug: Eldecalcitol capsules
- Calcitriol (Active Comparator): Participants receive oral calcitriol 0.5μg daily for 12 months
  Interventions: Drug: Calcitriol capsules

INTERVENTIONS:
Drug: Eldecalcitol capsules — Oral eldecalcitol 0.75μg daily
  Other Names: Edirol
  Arms: Eldecalcitol
Drug: Calcitriol capsules — Oral calcitriol 0.5μg daily
  Other Names: Haidewei
  Arms: Calcitriol

SUMMARY:
To investigate the efficacy and safety of eldecalcitol in postmenopausal women with low bone mineral density (BMD) or mild osteoporosis through a randomized, open-label, parallel controlled trial with calcitriol as the control.

DETAILED DESCRIPTION:
Postmenopausal women with low bone mineral density (BMD) or mild osteoporosis will be randomized in a 1:1 ratio to receive open-label oral 0.75μg eldecalcit daily or open-label oral 0.5μg calcitriol daily for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (based on medical history) aged 50 or older and menopause time more than 2 years. If there is uncertainty regarding menopausal status, women 60 years of age and older will be considered postmenopausal.
2. BMD (determined by DXA) of lumbar L1-4 or total hip or femoral neck met one of the following conditions at screening:

1) low BMD: -2.5<T< -1.0, without vertebral and fragility fracture history 2) mild osteoporosis: T≤-2.5, without vertebral and fragility fracture history 3. Ambulatory outpatients 4. Written informed consent

Exclusion Criteria:

1. Severe vitamin D deficiency at screening (defined as serum 25OHD<10 ng/ml);Vitamin D repletion will be permitted and dosage will be at the discretion of investigators and subjects may be re-screened
2. Primary hyperparathyroidism, Cushing's syndrome, hyperthyroidism, gonadal insufficiency, osteogenesis impotence, rheumatoid arthritis, poorly controlled diabetes mellitus (HbA1c>9%), or other conditions that can cause secondary osteoporosis, or treatment with glucocorticoids in the 2 months prior to study entry
3. Had injected bisphosphonate once or more within 3 years before entering the study; or had received oral bisphosphonate oral for 6 months or more in the 3 years prior to study entry; or had received parathyroid hormone once or more in the 3 years before entering the study; or received 2 weeks or more of calcitonin or vitamin K or active vitamin D or selective estrogen receptor modulator or hormone replacement therapy or traditional Chinese medicine for bone pine within 2 months prior to study entry; or received subcutaneous anti-RANKL antibody at any time prior to study entry
4. Urolithiasis at screening
5. Hypercalcemia (serum calcium >10.4 mg/dL), or hypercalciuria (urine calcium>400 mg/gCr), or hyperuricemia (above 420 μmol/L in men and 360 μmol/L in women)
6. Severe liver disease such as cirrhosis or serious heart disease such as severe heart failure
7. Active malignant tumors or a history of malignant tumors within 5 years before informed consent obtained
8. History of allergy to vitamin D
9. Any condition which in the opinion of the investigator unfit for the study

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline at Month 12 in BMD at the Lumbar Spine | Baseline to 12 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.

SECONDARY OUTCOMES:
Percent Change From Baseline at Month 6 in BMD at the Lumbar Spine | Baseline to 6 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.
Percent Change From Baseline at Month 6 in BMD of the Total Hip | Baseline to 6 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.
Percent Change From Baseline at Month 6 in BMD of the Femoral Neck | Baseline to 6 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.
Percent Change From Baseline at Month 12 in BMD of the Total Hip | Baseline to 6 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.
Percent Change From Baseline at Month 12 in BMD of the Femoral Neck | Baseline to 12 months
  Bone mineral density will be measured using dual energy x-ray absorptiometry (DXA). Images will be analyzed by a central imaging reader.
Percent Change From Baseline in Procollagen Type 1 N-telopeptide (P1NP) | Baseline and months 6 and 12
  Serum P1NP will be determined
Percent Change From Baseline in Type 1 Collagen C-telopeptide (CTX) | Baseline and months 6 and 12
  Serum CTX will be determined
Percent Change From Baseline in Parathyroid Hormone (PTH) | Baseline and months 6 and 12
  Serum PTH will be determined
Percent Change From Baseline in 25-Hydroxyvitamin D [25(OH)D] | Baseline and months 6 and 12
  Serum 25(OH)D will be determined
Incidence of new vertebral fracture | Baseline and months 12
  New vertebral fracture will be confirmed by the lateral X-ray of thoracic/lumbar vertebrae

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlin Zhang, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (21):
- China (21):
  - The Second Xiangya Hospital of Central South University, Changsha
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Ha’erbin
  - Huai 'an First People's Hospital, Huai'an
  - Liaocheng People's Hospital, Liaocheng
  - Jiangxi Provincial People's Hospital, Nanchang
  - Jiangsu Geriatric Hospital, Nanjin
  - The First Hospital of Ningbo, Ningbo
  - The Sixth Hospital of Ningbo, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Pudong New Area Punan Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Zhongshan Hosiptal Affiliated to Fudan University, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - The First Hospital of Shanxi Medical University, Taiyuan
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Hospital, Tianjin
  - Xi'an Honghui Hospital, Xi'an
  - Xuzhou Central Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: No